CLINICAL TRIAL: NCT06582368
Title: Determinants of Portal Vein Pulsatility Index: An Observational Study
Brief Title: Determinants of Portal Vein Pulsatility Index
Status: Completed | Type: Observational
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Principal Investigator, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Other Study IDs: 9593/04.04.2024
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fluid Overload; Congestion
Keywords: congestion; portal vein pulsatility; fluid therapy; right ventricular failure; volemia
MeSH Terms: conditions — Edema; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Mechanically ventilated postoperative adult patients after cardiac surgery within 6 hours after intensive care unit admission.

SUMMARY:
The pulsatile pattern of the portal vein is considered a marker of right ventricular dysfunction, but volemia may also contribute to this phenomenon. The separate influence of each factor remains debated, as the interplay between right ventricular dysfunction and volume status is complex. Additionally, right ventricular dysfunction can originate from either diastolic or systolic dysfunction, further complicating the understanding of their distinct impacts on portal vein pulsatility.

DETAILED DESCRIPTION:
The pulsatile pattern of the portal vein has been recognized as a potential marker of right ventricular dysfunction, reflecting altered hemodynamics in the venous system. However, the role of volemia, or the volume status of a patient, might also significantly influence this pulsatility, complicating the interpretation of portal vein flow patterns. The distinct and combined effects of right ventricular dysfunction and volemia on portal vein pulsatility are still subjects of ongoing debate. Right ventricular dysfunction itself can arise from multiple mechanisms, including primary diastolic dysfunction, where the ventricle has impaired filling and relaxation, or systolic dysfunction, characterized by reduced contractility and ejection capacity. Understanding whether diastolic or systolic dysfunction plays a predominant role in altering portal vein pulsatility is crucial, as these nuances have important implications for accurately identifying the determinants of portal vein pulsatility index and tailoring appropriate clinical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Mechanically ventilated patients within 6 hours after ICU admission following surgery who are considered for fluid administration to optimize haemodynamics.
* Sinus rhythm.

Exclusion Criteria:

* A condition known to interfere with portal vein flow assessment or interpretation (liver cirrhosis or chronic hepatic disease, suprahepatic or portal vein thrombosis).
* Any mechanical circulatory support.
* Cardiac transplant.
* Poor transthoracic echocardiographic window.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated postoperative adult patients after cardiac surgery within 6 hours after intensive care unit admission.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Fluid Intolerance | Within the first six hours of admission to the intensive care unit (simultaneously with other measures).
  A portal vein pulsatility index greater than 50%, calculated as (Vmax - Vmin) / Vmax, with no upper limit and 0% as the minimum limit. Higher values indicate worse outcomes. Ultrasonographic portal spectral waveform was used to measure Vmax and Vmin.

SECONDARY OUTCOMES:
Volemia | Within the first six hours of admission to the intensive care unit (simultaneously with other measures).
  Volemia will be assessed using the mean systemic filling pressure analogue (MSFPa) proposed by Parkin and Leaning (2008), which estimates the overall volume status and preload of the circulatory system. This measurement provides an indirect evaluation of volemia, reflecting the balance between blood volume and vascular capacity. Higher or lower values can indicate fluid overload or deficit, respectively.
Right Ventricular Dysfunction | Within the first six hours of admission to the intensive care unit (simultaneously with other measures).
  Right ventricular dysfunction will be assessed using three ancillary measures: Tricuspid Annular Plane Systolic Excursion (TAPSE), Right Ventricular Fractional Area Change (RVFAC), and the Right Ventricular End-Diastolic Area to Left Ventricular End-Diastolic Area ratio (RVEDA/LVEDA). TAPSE measures longitudinal shortening of the right ventricle, RVFAC assesses overall systolic function by evaluating the change in the right ventricular area during the cardiac cycle, and RVEDA/LVEDA compares the size of the right ventricle to the left, indicating potential dilation or pressure overload.

CONTACTS AND LOCATIONS:
Overall Officials: Serban-Ion Bubenek-Turconi, Professor, Study Director — "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases
Locations (1):
- "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases, Bucharest, Romania

REFERENCES:
- [Background] Parkin WG, Leaning MS. Therapeutic control of the circulation. J Clin Monit Comput. 2008 Dec;22(6):391-400. doi: 10.1007/s10877-008-9147-7. Epub 2008 Nov 12. PMID 19002596
- [Background] Utrilla-Alvarez JD, Gopar-Nieto R, Garcia-Cruz E, Lazcano-Diaz E, Jimenez-Rodriguez GM, Rojas-Velasco G, Manzur-Sandoval D. Assessing the venous system: Correlation of mean systemic filling pressure with the venous excess ultrasound grading system in cardiac surgery. Echocardiography. 2023 Nov;40(11):1216-1226. doi: 10.1111/echo.15697. Epub 2023 Sep 23. PMID 37742087